CLINICAL TRIAL: NCT05602168
Title: Collection of Sequential Samples From Patients With Malignant Myeloid Hemopathy for the Study of Treatment Resistance: HEMATOBIO.02-IPC 2021-061
Brief Title: Collection of Sequential Samples From Patients With Malignant Myeloid Hemopathy for the Study of Treatment Resistance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEMATOBIO.02-IPC 2021-061
Record Dates: First submitted 2022-10-10; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Hematologic Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: the study is interventional because there are blood samples taken outside the scope of routine care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental:Acute leukemia/myelodysplastic or myeloproliferative disease (Experimental): blood sampling, bone marrow aspirate, and buccal swab
  Interventions: Other: experimental:Acute leukemia/myelodysplastic or myeloproliferative disease

INTERVENTIONS:
Other: experimental:Acute leukemia/myelodysplastic or myeloproliferative disease — blood sampling, bone marrow aspirate and buccal swab

SUMMARY:
The main objective is to study the genomic, transcriptomic, proteomic epigenomic, metabolomic and immune mechanisms of blasts and microenvironment cells associated with IT resistance through the constitution of a collection associating blood or marrow samples from patients with LA, MDS and MPS marrow samples from patients with LA, MDS and MPS at diagnosis, during treatment and at relapse and relapse and clinical annotations.

DETAILED DESCRIPTION:
It is a collection of blood, marrow and oral epithelial cell samples taken longitudinally and oral epithelial cells taken longitudinally for each patient included, with each patient included, with the corresponding clinical data. An oral epithelial cell sample will be collected at inclusion from 2 swabs, which will allow extraction of DNA from healthy from healthy cells. During blood sampling necessary for care, an additional 40 ml of blood will be collected of 40 ml of blood will be collected in 10 tubes of 4 ml: 4 EDTA tubes, 4 heparinized heparinized tubes and 2 dry tubes. These additional collections will take place at the following times:

* At inclusion
* 7 days (+/- 2 days) after initiation of treatment
* 14 days (+/- 2 days) after initiation of therapy
* 21-42 days after initiation of therapy (early response assessment)
* In case of complete remission
* In case of relapse or progression During bone marrow punctures required for treatment, 6 ml of bone marrow bone marrow will be collected in 2 tubes of 3 ml: 1 EDTA tube and 1 heparinized tube.

heparinized tube. These additional collections will take place at the following times following times:

* At inclusion
* 21-42 days after initiation of treatment (assessment of early response) early response)
* In case of complete remission
* In case of relapse or progression Patients will be followed for up to 2 years after inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute leukemia, myelodysplastic syndrome, chronic myelomonocytic leukemia (CMML) or myeloproliferative syndrome according to the WHO classification 2016,
2. Patient for whom a new line of therapy is initiated.
3. Patient older than 18 years of age.
4. Patient affiliated to the social security system or benefiting from such a system.
5. Signed consent to participate.

Exclusion Criteria:

1. Weight at inclusion < 50 kg
2. Participating in another clinical study that would cause the total amount of blood collection to exceed the and endanger the patient
3. Person in an emergency situation, adult under legal protection (guardianship, curatorship, etc.) protection (guardianship, curatorship or safeguard of justice), or unable to express his or her consent.
4. Impossibility to submit to the medical follow-up of the trial for geographical social or psychological reasons,
5. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Acute leukemia/ Myeloproliferative/ myelodysplastic syndrome cells profiling (molecular analysis, epigenetic profile, drug sensitivity profile,immunophenotyping) | up to 7 years
  establishment of genomic and proteomic signatures as well as transcriptomic and metabolic profiles associated with IT resistance.

SECONDARY OUTCOMES:
to study the resistance to treatments | up to 7 years
  study of the sensitivity to IT in vitro of primary cells from patients
Creation of murine cell models (Patient-derived xenografts, PDX) from patient blasts to study in vivo in order to study in vivo the mechanisms of resistance to treatment. | up to 7 years
  Establishment of xenografts in immunocompromised mice from primary cells of TI-resistant patients patients resistant to IT